CLINICAL TRIAL: NCT00090831
Title: Investigating the Role of Serotonin in Emotional Processing Through the Use of Tryptophan Depletion
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040270; 04-M-0270
Record Dates: First submitted 2004-09-03; First posted 2004-09-06 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2012-09-17

CONDITIONS: Healthy
Keywords: Emotional Learning; Neurotransmitter; Neural Systems; Response Control; Orbitofrontal Cortex; Amygdala; Serotonin; Healthy Volunteer; HV

SUMMARY:
This study will examine the role of serotonin function in the brain. Serotonin, one of the brain's natural chemicals, connects with receptors on brain cells to regulate emotion, anxiety, sleep, stress hormones, and other body functions that are disturbed in various mood and anxiety disorders. Also, the research will look at the function of particular brain areas, how they are involved in regulating emotions, and how serotonin is involved in the regulation of their function. The procedures entailed are tryptophan depletion and magnetic resonance imagining (MRI). Also, researchers' understanding of the genetic causes of mood and anxiety disorders will increase through examination of participants' DNA.

Adults in good health, ages 20 through 50, may be eligible for this study. Among those not eligible are females who are pregnant or breast feeding, patients with psychiatric or central nervous system disease, and those taking medications that would interfere with study results.

At the first visit, patients will be asked about their general mood, degree of nervousness, thinking skills, and behavior. The session will last from 1.5 to 2.0 hours. A blood sample of about 2 tablespoons will be drawn, for DNA study.

Participants will undergo the following procedures and tests:

* Physical examination.
* Test of vital signs, lying and standing.
* Electrocardiogram.
* Collection of blood for chemistry and hematology.
* Urinalysis.
* HIV, urine drug, and hepatitis screening.
* Psychiatric screening.
* (SqrRoot) -HCG pregnancy test, if applicable.

At the second visit, patients will receive either tryptophan depletion or placebo, and 5 hours later, the study will begin, to last up to 2 additional hours. Patients will be asked periodically about their emotional state or changes in their well-being. The MRI system will create images of the brain's blood flow and measure glucose metabolism as a measure of brain activity. During the MRI scan, patients will hear knocking or beeping sounds, and they will wear earplugs to reduce the noise. Patients will be able to communicate with the MRI staff at all times during the scan, and they may ask to be moved out of the machine at any time. The MRI session lasts up to 1.5 hours.

Results of any medical tests or other information will not be provided to participants, because further research may be needed before such results are meaningful. But if meaningful information develops from this study that may be important for a participant's health, he or she will be notified about it when it becomes available.

DETAILED DESCRIPTION:
Objective

The goal of this protocol is to use a targeted serotonergic manipulation [acute tryptophan depletion (ATD)] and specific neurocognitive and neuroimaging paradigms to consider the role of serotonin (5-HT) in emotional processing. In particular, we wish to evaluate claims that serotonin has a role in the effective processing of aversive signals. Additionally, we wish to examine whether tryptophan depletion will attenuate the neural response to aversive material.

Study population

Healthy human adult volunteers, ages 20-50 years old, with no DSM-IV-defined Axis I mental disease and who fulfill the remainder of the inclusion/exclusion criteria.

Design

This is a prospective, randomized, double-blind, placebo-controlled, single-dose, outpatient study in eligible, healthy volunteers. Participants will be randomly assigned in a 1:1 ratio to single doses of drug (ATD) or placebo. The National Institutes of Health (NIH) Clinical Center Pharmacy will facilitate randomization and supply the randomization code to the Clinical Center s Metabolic Nutrition Department (see below). All subjects will be monitored for adverse events. Participants will give written, informed consent prior to any assessments and procedures covered by this protocol.

The study will be conducted in the NIH Clinical Center 5SW Day Hospital and the NMRF center (for the imaging arm of the study). Subjects will arrive in the morning of the testing day and complete baseline measurements (i.e., mood and anxiety ratings and serum tryptophan levels). Participants will then receive an oral dose of ATD capsules or placebo. Participants will consume two meals during the study day; the placebo group (control subjects) will be given high-tryptophan meals and tryptophan-depleted subjects will receive low-tryptophan meals. Meals will be designed and supplied by the NIH Clinical Center Metabolic Nutrition Department. At specified times, subjects will complete primary measures [either neurocognitive or neuroimaging (fMRI) paradigms] and secondary measures (mood and anxiety ratings and serum levels of tryptophan) as detailed in the protocol. Adverse events will be monitored throughout the study day. A post-study evaluation will occur prior to discharging the participant to verify that he/she is physically and mentally well and fit to leave the Clinical Center.

Outcome Measures

Primary Outcome Measures:

* Neurocognitive Paradigms: Behavioral measures including reaction time and accuracy
* Neuroimaging Paradigms: Blood-oxygen-level-dependent (BOLD) response

Secondary Outcome Measurements:

* Serum tryptophan levels
* Mood and Anxiety Rating Scales

ELIGIBILITY:
* INCLUSION CRITERIA:

Age: Participants will be males and females, 20-50 years of age.

IQ: IQ, as measured by 4 subscales from the Wechsler Adult Intelligence Scale-Revised (WAIS-R), must be greater than 80.

Participants will be able to comprehend the purpose and procedures of the study. They will be able to provide written, informed consent for all study procedures.

EXCLUSION CRITERIA:

Psychiatric history: Participants will be assessed using DSM-IV criteria via standardized psychiatric interviews conducted by trained examiners (SCID). All participants will be free of any current or past major affective disorder, psychotic disorder, substance dependence, anorexia nervosa or bulimia. All participants will be free of any current anxiety disorders with the exception of specific phobias and free of current somatoform disorders. In addition, participants with a first degree relative with major depressive disorder will be excluded.

Severe acute and chronic medical illnesses (e.g., cardiac disease, diabetes, epilepsy).

CNS disease: History of brain abnormalities (e.g., neoplasms, subarachnoid cysts), cerebrovascular disease, infectious disease (e.g., abscess), or other neurological disease, or history of head trauma (defined as loss of consciousness greater than 3 min).

Currently on any regular medication that would interfere with study results (with exception of contraceptive pill).

Current use of psychotropic medication or benzodiazepine

Currently breast feeding or pregnant (as documented by pregnancy testing done within 24 hr of the study starting)

Subjects who are lactose intolerant will be excluded as the placebo capsules contain lactose. Also, those subjects who cannot consume the diets provided by metabolic nutrition on the study day will be excluded.

ADDITIONAL EXCLUSION CRITERIA FOR fMRI STUDIES:

Metal or electronic objects: Metal plates, certain types of dental braces, cardiac pacemakers, etc., that are sensitive to electromagnetic fields contraindicate MRI scans.

Claustrophobia: participants will be questioned about potential discomfort in being in an enclosed space, such as an MRI scanner.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2004-08-31; Study Completion 2012-09-17

CONTACTS AND LOCATIONS:
Overall Officials: James J Blair, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abbott FV, Etienne P, Franklin KB, Morgan MJ, Sewitch MJ, Young SN. Acute tryptophan depletion blocks morphine analgesia in the cold-pressor test in humans. Psychopharmacology (Berl). 1992;108(1-2):60-6. doi: 10.1007/BF02245286. PMID 1410147
- [Background] Adolphs R. Neural systems for recognizing emotion. Curr Opin Neurobiol. 2002 Apr;12(2):169-77. doi: 10.1016/s0959-4388(02)00301-x. PMID 12015233
- [Background] Aron AR, Fletcher PC, Bullmore ET, Sahakian BJ, Robbins TW. Stop-signal inhibition disrupted by damage to right inferior frontal gyrus in humans. Nat Neurosci. 2003 Feb;6(2):115-6. doi: 10.1038/nn1003. No abstract available. PMID 12536210